CLINICAL TRIAL: NCT01363037
Title: Phase 1 Safety and Pharmacokinetics of Dapivirine/Maraviroc Vaginal Ring
Brief Title: Safety and Pharmacokinetics of Dapivirine/Maraviroc Vaginal Ring
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: International Partnership for Microbicides, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MTN-013/IPM 026
Record Dates: First submitted 2011-05-27; First posted 2011-06-01 (Estimated); Last update posted 2015-09-10 (Estimated); Status verified 2015-09

CONDITIONS: HIV Infections
Keywords: HIV infections; Anti-HIV agents; HIV-1
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Dapivirine-Maraviroc Vaginal Ring (Experimental)
  Interventions: Drug: Dapivirine-Maraviroc Vaginal Ring
- Placebo Vaginal Ring (Placebo Comparator)
  Interventions: Other: Placebo Vaginal Ring
- Maraviroc Vaginal Ring (Active Comparator)
  Interventions: Drug: Maraviroc Vaginal Ring
- Dapivirine Vaginal Ring (Active Comparator)
  Interventions: Drug: Dapivirine Vaginal Ring

INTERVENTIONS:
Drug: Dapivirine Vaginal Ring — dosage form: dapivirine vaginal ring dosage:25 mg frequency:continuous use duration:28 days
  Arms: Dapivirine Vaginal Ring
Drug: Maraviroc Vaginal Ring — dosage form: maraviroc vaginal ring dosage:100 mg frequency:continuous use duration:28 days
  Arms: Maraviroc Vaginal Ring
Other: Placebo Vaginal Ring — dosage form: placebo vaginal ring dosage:N/A frequency:continuous use duration:28 days
  Arms: Placebo Vaginal Ring
Drug: Dapivirine-Maraviroc Vaginal Ring — dosage form: combination vaginal ring dosage:25 mg dapivirine + 100 mg maraviroc frequency:continuous use duration:28 days
  Arms: Dapivirine-Maraviroc Vaginal Ring

SUMMARY:
The purpose of this study is to assess the pharmacokinetics of the combination dapivirine and maraviroc vaginal ring and determine whether it is safe when used continuously for 28 days by healthy women in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 through 40 years (inclusive) at screening, verified per site SOPs
* Able and willing to provide written informed consent to be screened for and take part in the study
* Able and willing to provide adequate locator information, as defined by the site SOPs
* HIV-uninfected, based on testing performed by study staff at Screening and Enrollment (per applicable algorithm in Appendix II)
* In general good health at Screening and Enrollment, as determined by the site IoR or designee
* At Screening, participant states willingness to abstain from receptive sexual activity (including oral, vaginal and anal intercourse) for the 14 days prior to enrollment and for the duration of study participation
* Per participant report, using an effective method of contraception at Enrollment, and intending to continue use of an effective method for the duration of study participation. Effective methods include hormonal methods (except contraceptive vaginal rings), intrauterine device (IUD) inserted at least 28 days prior to enrollment, being a woman who identifies as a woman who has sex with women exclusively, sterilization, and/or sexually abstinent for the past 90 days
* Satisfactory Pap result in the 12 calendar months prior to Enrollment consistent with Grade 0 according to the Female Genital Grading Table for Use in Microbicide Studies Addendum 1 to the DAIDS Table for Grading Adult and Pediatric Adverse Events, Version 1.0, December 2004 (Clarification dated August 2009), or satisfactory evaluation with no treatment required of Grade 1 or higher Pap result per American Society for Colposcopy and Cervical Pathology (ASCCP) guidelines in the 12 calendar months prior to Enrollment.
* Per participant report at Screening and Enrollment, agrees not to participate in other research studies involving drugs, medical devices, or vaginal products for the duration of study participation
* Per participant report at Screening, regular menstrual cycles with at least 21 days between menses (does not apply to participants who report using a progestin-only method of contraception at screening, e.g., Depo-Provera or levonorgestrel-releasing IUD)
* At Screening and Enrollment, participant states a willingness to refrain from inserting any non-study vaginal products or objects into the vagina, including but not limited to, spermicides, female condoms, diaphragms, contraceptive vaginal rings, vaginal medications, menstrual cups, cervical caps (or any other vaginal barrier method), douches, lubricants, sex toys (vibrators, dildos, etc.), and tampons for the 5 days prior to enrollment throughout the duration of study participation. -- Note: At the Screening visit participant also agrees to refrain from the practices listed above for at least 5 days prior to enrollment.

Exclusion Criteria:

* Participant report of any of the following at Screening:

  * Known adverse reaction to silicone, titanium dioxide, or to any of the components of the study products
  * Use and/or anticipated use during the period of study participation of CYP3A inducer(s) and/or inhibitor(s)
  * Chronic and/or recurrent candidiasis
  * Non-therapeutic injection drug use in the 12 months prior to screening
  * Post-exposure prophylaxis for HIV exposure within 6 months prior to screening
  * Last pregnancy outcome 90 days or less prior to screening
  * Currently breastfeeding
  * Hysterectomy
  * Intends to become pregnant within the next 4 months
  * Has plans to relocate away from the study site area in the next 4 months
* Reports participating in any other research study involving drugs, medical devices, or vaginal products 60 days or less prior to enrollment
* At Screening or Enrollment, as determined by the IoR/designee, any significant uncontrolled active or chronic cardiovascular, renal, liver, hematologic, neurologic, gastrointestinal, psychiatric, endocrine, respiratory, immunologic disorder or infectious disease, or at increased risk of cardiovascular events
* Has any of the following laboratory abnormalities at Screening:

  * Aspartate aminotransferase (AST) or alanine transaminase (ALT) Grade 1 or higher as per the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events Version 1.0, December, 2004 (Clarification dated August 2009)
  * Calculated creatinine clearance less than 60 mL/min by the Cockcroft- Gault formula, where creatinine clearance (female) in mL/min = (140 - age in years) x (weight in kg) x (0.85)/72 x (creatinine in mg/dL)
  * Hemoglobin Grade 1 or higher as per the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events Version 1.0, December, 2004 (Clarification dated August 2009)
  * Platelet count Grade 1 or higher as per the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events Version 1.0, December, 2004 (Clarification dated August 2009) --- Note: Otherwise eligible participants with an exclusionary test result may be retested during the screening process. If a participant is re- tested and a nonexclusionary result is documented within 45 days of providing informed consent for screening, the participant may be enrolled.
* At Screening or Enrollment, is pregnant
* Diagnosed with urinary tract infection (UTI) at Screening or Enrollment

  -- Note: Otherwise eligible participants diagnosed with UTI during screening will be offered treatment and may be enrolled after completing treatment and all symptoms have resolved. If treatment is completed and symptoms have resolved within 45 days of obtaining informed consent for screening, the participant may be enrolled.
* Diagnosed with pelvic inflammatory disease, a sexually transmitted infection (STI) or reproductive tract infection (RTI) requiring treatment per current Centers for Disease Control and Prevention (CDC) guidelines (http://www.cdc.gov/std/treatment/) at Screening or Enrollment

  -- Note: Otherwise eligible participants diagnosed with STI or RTI during screening will be offered treatment and may be enrolled after completing treatment and all symptoms have resolved. If treatment is completed and symptoms have resolved within 45 days of obtaining informed consent for screening, the participant may be enrolled.
* At Screening or Enrollment, has a clinically apparent Grade 1 or higher pelvic exam finding (observed by study clinician or designee) per the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 1.0, December 2004 (Clarification dated August 2009), Addendum 1, Female Genital Grading Table for Use in Microbicide Studies

  -- Note: Cervical friability bleeding associated with speculum insertion and/or specimen collection judged to be within the range of normal according to the clinical judgment of the IoR/designee is considered expected non-menstrual bleeding and is not exclusionary.
* At Screening, severe pelvic relaxation such that either the vaginal walls or the uterine cervix descend beyond the vaginal introitus with valsalva maneuver
* Has any other condition that, in the opinion of the IoR/designee, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving study objectives.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2011-11; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Safety: To assess and compare safety of VRs containing 25 mg dpv, or 100 mg mrv, or 25 mg dpv + 100 mg mrv, the endpoint was the proportion of women in the four arms experiencing specific, protocol defined safety events during the study (see description) | 7.5 weeks
  * Genitourinary events Grade 1 or higher as defined by the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 1.0, Dec 2004 (Clarification dated August 2009), Addendum 1, (Female Genital Grading Table for Use in Microbicide Studies) judged to be related to study product
  * Adverse events Grade 2 or higher as defined by the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 1.0, Dec 2004 (Clarification dated August 2009)
Pharmacokinetics: Assessments of systemic and local concentrations of dapivirine and maraviroc in plasma, vaginal fluids and cervical tissue, respectively | 7.5 weeks
  Assessed during and after 28 days' of continuous use of a vaginal ring containing 25 mg dapivirine, or 100 mg maraviroc, or 25 mg dapivirine + 100 mg maraviroc.

SECONDARY OUTCOMES:
Evaluate the acceptability of the study VR in HIV-uninfected sexually abstinent women over 28 days of use | 28 days
  Participant report of acceptability including genitourinary and emotional (dis)comfort, awareness/feeling during daily activities, ring insertion/removal issues, and willingness to use in the future
Evaluate the adherence to the study VR in HIV-uninfected sexually abstinent women over 28 days of use | 28 days
  Participant report of frequency of study VR removal/expulsions (voluntary and involuntary) and duration without VR inserted in vagina

CONTACTS AND LOCATIONS:
Overall Officials: Beatrice A Chen, MD, MPH, Study Chair — University of Pittsburgh; Lori Panther, MD, MPH, Study Chair — The Fenway Institute
Locations (3):
- United States (3):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - The Fenway Institute/Fenway Community Health, Boston, Massachusetts
  - Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Chen BA, Panther L, Marzinke MA, Hendrix CW, Hoesley CJ, van der Straten A, Husnik MJ, Soto-Torres L, Nel A, Johnson S, Richardson-Harman N, Rabe LK, Dezzutti CS. Phase 1 Safety, Pharmacokinetics, and Pharmacodynamics of Dapivirine and Maraviroc Vaginal Rings: A Double-Blind Randomized Trial. J Acquir Immune Defic Syndr. 2015 Nov 1;70(3):242-9. doi: 10.1097/QAI.0000000000000702. PMID 26034880